CLINICAL TRIAL: NCT07040033
Title: Investigation of the Relationship Between Strengthening and Ikigai Levels of Individuals With Coronary Artery Disease
Status: Recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Other Study IDs: KutahyaHSU20250525
Record Dates: First submitted 2025-06-11; First posted 2025-06-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-06

CONDITIONS: Coronary Arterial Disease (CAD); NURSİNG; Disease Management; LIFE SATISFACTION
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There will be no intervention — There will be no intervention
Behavioral: There will be no intervention — There will be no intervention

SUMMARY:
cardiac rehabilitation includes topics such as smoking cessation recommendations, weight management, nutritional counseling, blood pressure management, physical activity counseling, diabetes management, psychosocial management in order to reduce CV risk factors, reduce morbidity and mortality rates, and improve the individual's quality of life . In CV diseases, it has been shown that education and motivation provided under the leadership of nurses are effective in preventing the disease. This success stems from the nurse's holistic approach to the individual and determination of individual-specific needs. It is important for nurses, who are seen as a source of support by the society, to identify empowerment in CV patients and to support patients for independent living. kigai is a well-known term in Japan. This term is sometimes translated as 'purpose in life' and sometimes it can be defined as 'joy of life'. When Ikigai is mentioned, both the source of Ikigai within the individual or the object of Ikigai, and the psychological/emotional state (Ikigai-kan) in which Ikigai is felt come to mind. Accordingly, 'Ikigai' can be defined as the source or object of the purpose/joy of life, and 'Ikigai-kan' as the psychological/emotional state in which these are felt. In addition to the ways in which individuals with cardiovascular disease manage their disease, take precautions against risk factors, and perform strengthening exercises, determining the patients' current state of mind is also an important element. In this sense, physicians and nurses in the clinic take these elements into consideration when planning the care to be provided to patients.

No study has been found in the literature to date that evaluates the relationship between CAH strengthening and Ikigia. Based on this information, this study aims to examine the relationship between CAH strengthening and Ikigai.

It is expected that the research results will guide physicians and nurses who care for individuals with CAH in planning the care to be provided to patients and contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Coronary Artery Disease
* Must be in a stable phase of the disease
* Speak and understand Turkish
* Must be 18 years of age or older

Exclusion Criteria:

* Diagnosed with a mental illness or communication disorder
* Presence of significant hearing or vision disorders
* Intubated Coronary Artery Disease patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Title: Determining the relationship between empowerment and ikigai levels in individuals diagnosed with Chronic Lung Disease (CLD) | 2 months from the start of the study
  Description: The relationship between participants' empowerment levels and their ikigai levels will be evaluated using validated and reliable scales through descriptive statistics and correlation analysis.

SECONDARY OUTCOMES:
Relationship between sociodemographic characteristics and empowerment and ikigai levels | 2 months from the start of the study
  Description: Evaluation of the impact of variables such as age, gender, education level, and disease duration on empowerment and ikigai levels
Title: Relationship between quality of life and ikigai levels | 2 months from the start of the study
  Description: Determining whether there is a significant correlation between participants' quality of life and their ikigai levels

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Merkez, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No